CLINICAL TRIAL: NCT00156819
Title: The Leukotriene Modifier Or Corticosteroid or Corticosteroid-Salmeterol Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: JHSPH Center for Clinical Trials (Other)
Collaborators: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALAACRC-03
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Results first posted 2015-12-09 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-11

CONDITIONS: Asthma
Keywords: Asthma; Asthma Control
MeSH Terms: conditions — Asthma | interventions — Fluticasone; montelukast; Salmeterol Xinafoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Fluticasone (Active Comparator): Participants continued fluticasone (100 microgram twice daily) treatment.
  Interventions: Drug: fluticasone; Drug: montelukast; Drug: Fluticasone plus salmeterol
- Montelukast (Experimental): Participants were changed to Montelukast (5 or 10 mg each night).
  Interventions: Drug: fluticasone; Drug: montelukast; Drug: Fluticasone plus salmeterol
- Fluticasone plus salmeterol (Experimental): Participants were given fluticasone (100 microgram) plus salmeterol (50 microgram) each night.
  Interventions: Drug: fluticasone; Drug: montelukast; Drug: Fluticasone plus salmeterol

INTERVENTIONS:
Drug: fluticasone — fluticasone (100 microgram twice daily) treatment
Drug: montelukast — Montelukast (5 or 10 mg each night).
Drug: Fluticasone plus salmeterol — fluticasone (100 microgram) plus salmeterol (50 microgram) each night

SUMMARY:
This research study will compare the treatment effects of three different asthma medications in asthma subjects whose asthma is well controlled when they take fluticasone, an inhaled corticosteroid. The treatments are fluticasone, montelukast (an anti?leukotriene drug), and a combination therapy of fluticasone and salmeterol (a long-acting beta-agonist). Fluticasone, montelukast, and the combination therapy of fluticasone and salmeterol (Advair Diskus®) are all approved for the treatment of asthma. We are looking at whether the three treatments are equally effective for reducing the number and the severity of asthma attacks in subjects with mild to moderately severe asthma.

DETAILED DESCRIPTION:
This trial will attempt to investigate whether asthmatic patients that are well controlled with low-dose twice daily inhaled corticosteroid (ICS) therapy can safely be switched to other modes of controller therapy without loss of asthma control. Patients demonstrating good control on twice-daily low-dose ICS will be randomized to one of three treatment groups: once-daily low-dose ICS (fluticasone), leukotriene receptor antagonist (montelukast), or once-daily combination therapy (fluticasone-salmeterol).

ELIGIBILITY:
Inclusion Criteria:

* physician-diagnosed asthma
* age 6 or older
* pre-bronchodilator forced expiratory volume (FEV1) of at least 60% of predicted
* beta-agonist reversibility OR airways hyperreactivity by methacholine challenge
* Juniper Asthma Control Score of 1.5 or greater if not on daily controller
* good current health

Exclusion Criteria:

* current or past smoking (greater than 20 pack-years)
* chronic or current oral steroid therapy
* pregnancy, lack of effective contraception (when appropriate), lactation

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2003-06; Primary Completion 2005-08 (Actual); Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Anthonisen, MD, Study Chair — University of Winnipeg
Locations (19):
- United States (19):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - National Jewish Hospital, Denver, Colorado
  - Nemour's Childrens Center, Jacksonville, Florida
  - University of Miami (and University of South Florida in Tampa), Miami, Florida
  - Emory University, Atlanta, Georgia
  - Illinois Consortium (Northwestern, Univ. of Chicago, Univ. of Illinois), Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Louisiana State University, New Orleans, Louisiana
  - University of Minnesota, Minneapolis, Minnesota
  - University of Missouri at Kansas City, Kansas City, Missouri
  - Washington University, St Louis, Missouri
  - Long Island Jewish Hospital (and North Shore Hospital), New Hyde Park, New York
  - New York Consortium (New York Univ. and Columbia Univ.), New York, New York
  - New York Medical College, Valhalla, New York
  - Duke University School of Medicine, Durham, North Carolina
  - Ohio State University, Columbus, Ohio
  - Thomas Jefferson Hospital, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - Northern New England Consortium (Univ. of Vermont and other locations), Burlington, Vermont

REFERENCES:
- [Derived] Sharma R, Tiwari A, Kho AT, Wang AL, Srivastava U, Piparia S, Desai B, Wong R, Celedon JC, Peters SP, Smith LJ, Irvin CG, Castro M, Weiss ST, Tantisira KG, McGeachie MJ. Circulating microRNAs associated with bronchodilator response in childhood asthma. BMC Pulm Med. 2024 Nov 4;24(1):553. doi: 10.1186/s12890-024-03372-4. PMID 39497092
- [Derived] Sharma R, Tiwari A, Kho AT, Wang AL, Srivastava U, Piparia S, Desai B, Wong R, Celedon JC, Peters SP, Smith LJ, Irvin CG, Castro M, Weiss ST, Tantisira KG, McGeachie MJ. Circulating MicroRNAs associated with Bronchodilator Response in Childhood Asthma. Res Sq [Preprint]. 2023 Jun 29:rs.3.rs-3101724. doi: 10.21203/rs.3.rs-3101724/v1. PMID 37461659
- [Derived] Lang JE, Hossain J, Dixon AE, Shade D, Wise RA, Peters SP, Lima JJ; American Lung Association-Asthma Clinical Research Centers. Does age impact the obese asthma phenotype? Longitudinal asthma control, airway function, and airflow perception among mild persistent asthmatics. Chest. 2011 Dec;140(6):1524-1533. doi: 10.1378/chest.11-0675. Epub 2011 Jul 28. PMID 21799027
- [Derived] Duan QL, Gaume BR, Hawkins GA, Himes BE, Bleecker ER, Klanderman B, Irvin CG, Peters SP, Meyers DA, Hanrahan JP, Lima JJ, Litonjua AA, Tantisira KG, Liggett SB. Regulatory haplotypes in ARG1 are associated with altered bronchodilator response. Am J Respir Crit Care Med. 2011 Feb 15;183(4):449-54. doi: 10.1164/rccm.201005-0758OC. Epub 2010 Sep 17. PMID 20851928
- [Derived] American Lung Association Asthma Clinical Research Centers; Peters SP, Anthonisen N, Castro M, Holbrook JT, Irvin CG, Smith LJ, Wise RA. Randomized comparison of strategies for reducing treatment in mild persistent asthma. N Engl J Med. 2007 May 17;356(20):2027-39. doi: 10.1056/NEJMoa070013. PMID 17507702
- See also: American Lung Association Asthma Clinical Research Centers — http://www.cctrials.org/alaacrc

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fluticasone | Montelukast | Fluticasone Plus Salmeterol
Started | 169 | 166 | 165
Completed | 168 | 165 | 162
Not Completed | 1 | 1 | 3
Not completed — Lost to Follow-up | 1 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluticasone | Montelukast | Fluticasone Plus Salmeterol | Total
Number analyzed (Participants) | 169 | 166 | 165 | 500
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.3 (14.6) | 32.4 (15.4) | 30.8 (14.9) | 30.8 (15.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 95 | 103 | 301
  Male | 66 | 71 | 62 | 199

OUTCOME MEASURES:

1. Primary Outcome: Treatment Failure
Description: The primary outcome measure was treatment failure, defined as the occurrence of any one of the following events: hospitalization or an urgent medical visit for asthma initiated by the patient or physician; use of systemic corticosteroids for asthma or need for open-label use of inhaled corticosteroids for asthma, as determined by the study physician or an asthma care provider; a decrease in prebronchodilator forced expiratory volume in 1 second (FEV1) to more than 20% below the baseline value measured at randomization; a decrease in the morning peak expiratory flow rate to more than 35% below the baseline value (the mean over the final 2 weeks of the run-in period) on 2 consecutive days; use of 10 puffs or more per day of rescue beta-agonist for 2 consecutive days (except as medication before exercise); refusal of the patient to continue because of lack of satisfaction with treatment; or judgment by a physician that the patient should stop treatment for reasons of safety.
Time Frame: 16 weeks
Measure: Number; unit: participants
Arm/Group | Fluticasone | Montelukast | Fluticasone Plus Salmeterol
Number analyzed (Participants) | 168 | 165 | 162
participants | 34 | 50 | 33

ADVERSE EVENTS:
Arm/Group | Fluticasone | Montelukast | Fluticasone Plus Salmeterol
Serious Adverse Events (participants affected / at risk) | 6/168 | 4/165 | 4/162
Other Adverse Events (participants affected / at risk) | 159/168 | 156/165 | 157/162
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fluticasone (N=168) | Montelukast (N=165) | Fluticasone Plus Salmeterol (N=162)
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0 — Suffered concussion while snowboarding.
Chest pain (Cardiac disorders) | 1 | 0 | 0
Partial right knee replacement surgery (Surgical and medical procedures) | 1 | 0 | 0
Drop in peak flow (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Anaphylactic reaction to peanuts (Injury, poisoning and procedural complications) | 1 | 0 | 0
Asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1
Allergic reaction to Bactim (Injury, poisoning and procedural complications) | 0 | 0 | 1
Elbow sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Abcess (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tonsilectomy (Surgical and medical procedures) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fluticasone (N=168) | Montelukast (N=165) | Fluticasone Plus Salmeterol (N=162)
Upper respiratory infection (Infections and infestations) | 63 | 44 | 62
Pharyngitis (Infections and infestations) | 83 | 82 | 78
Rhinitis (Infections and infestations) | 120 | 111 | 118
Upper respiratory inflammation (Respiratory, thoracic and mediastinal disorders) | 84 | 67 | 73
Hoarsness/ dysphonia (General disorders) | 92 | 78 | 87
Sinisitis (Infections and infestations) | 67 | 51 | 50
Nasal congestion (General disorders) | 136 | 127 | 129
Viral respiratory infection (Infections and infestations) | 26 | 12 | 22
Influenza (Infections and infestations) | 15 | 8 | 16
Headache (General disorders) | 120 | 117 | 112
Diarrhea (General disorders) | 41 | 35 | 31
Nausea and vomitting (Gastrointestinal disorders) | 55 | 35 | 37
Gastrointestinal distress (Gastrointestinal disorders) | 63 | 57 | 61
Fever (Infections and infestations) | 45 | 25 | 36
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 63 | 71 | 70

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No